CLINICAL TRIAL: NCT03648060
Title: Efficacy of a Home-based Rehabilitation Program Performed Through a Digital Kinematic Biofeedback System After Total Hip or Knee Replacement: a Single-arm, Prospective, Open-label Study
Brief Title: Efficacy of a Digital Biofeedback System for Home-based Rehabilitation After Total Joint Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sword Health, SA (Industry)
Collaborators: Hospital da Prelada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH-SA-TJR-01
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-03

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Home-based rehabilitation sessions performed with the digital kinematic biofeedback system. Patients will be instructed to perform exercise sessions in at least 5 days per week, but compliance to this schedule is not mandatory per protocol.
  Interventions: Device: Digital kinematic biofeedback system

INTERVENTIONS:
Device: Digital kinematic biofeedback system — The system will be used independently by the patients to perform rehabilitation sessions at home, under remote monitoring from the clinical team. A tailored rehabilitation program will be prescribed by the therapist and edited according to patient evolution.
  Other Names: SWORD Phoenix

SUMMARY:
The study was designed to assess the efficacy of a home-based rehabilitation program using a digital kinematic biofeedback system after total hip or knee replacement.

This is a single-arm prospective study. Patients will be enrolled pre-operatively and will perform an 8-week rehabilitation program starting between day 7 and 10 after surgery.

This program will consist of rehabilitation sessions performed independently by the patient at under remote monitoring from a physical therapist.

Outcomes will be measured at baseline, 4 weeks into the rehabilitation program and at the end of the program.

The primary outcome is the change in patient performance measure through the Timed-up-and-Go (TUG) test in comparison with the pre-operative score. Secondary outcomes will be measured in terms of: a) patient reported outcomes (Hip or Knee Osteoarthritis Outcome Score) and b) range of motion of the relevant joint (hip or knee).

ELIGIBILITY:
Inclusion Criteria:

* Clinical and imaging evidence of hip/knee osteoarthritis
* Indication for total hip/knee replacement according to the patient´s orthopedic surgeon
* Ability to walk unaided, with unilateral or bilateral support
* Availability of a carer to assist the patient after surgery

Exclusion Criteria:

* Patients admitted for revision of total hip/knee replacement
* Contralateral hip or knee osteoarthritis severely limiting patient mobility and ability to comply with a rehabilitation program
* Aphasia, dementia or psychiatric comorbidity interfering with the communication or compliance to the rehabilitation process
* Respiratory, cardiac, metabolic or other condition incompatible with at least 30 minutes of light to moderate physical activity
* Major medical complications occurring after surgery that prevent the discharge of the patient within 10 days after the surgery
* Other medical and/or surgical complications that prevent the patient from complying with a rehabilitation program
* Blind and/or illiterate patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Change in the Timed up and Go Test score | Baseline, 4 weeks into the rehabilitation program and at the end of the program (week 8)
  The timed up and go requires a patient to rise from a chair walk three meters around a piece of tape and return to the chair again as quickly as possible.

SECONDARY OUTCOMES:
Change in the Hip Osteoarthritis Outcome Score/Knee Osteoarthritis Outcome Score | Baseline, 4 weeks into the rehabilitation program and at the end of the program (week 8)
  The HOOS/KOOS are standardized and validated patient outcome scores that assess functional limitation in patient with hip/knee osteoarthritis
Change in Hip/Knee Range of Motion | Baseline, 4 weeks into the rehabilitation program and at the end of the program (week 8)
  This will be measured (in degrees) automatically by the device

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, Principal Investigator — Sword Health, SA; Rosmaninho Seabra, MD, Study Chair — Hospital da Prelada
Locations (1):
- Hospital da Prelada, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Yes The study protocol will be made available in PDF format. Aggregate study results, with anonymised individual participant data will be made available in Excel format.
Supporting Information: Study Protocol, SAP
Time Frame: Upon study publication, for at least five years.
Access Criteria: Study protocol will be made available here and the excel file with the aggregate results will be made available upon study publication, for at least 5 years.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT03648060/Prot_SAP_001.pdf